CLINICAL TRIAL: NCT02828800
Title: Cartography of Allodynic and Hypoasthetic Territories Associated With Neuropathic Pain Following Total Knee Arthroplasty (TKA)
Brief Title: Cartography of Allodynic and Hypoasthetic Territories Following TKA
Acronym: CARTODOL
Status: Terminated | Type: Observational
Why Stopped: investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0034
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Pain, Postoperative; Neuropathic Pain
MeSH Terms: conditions — Pain, Postoperative; Neuralgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cartography of allodynic and hypoasthetic territories — The cartography of allodynic and hypoasthetic territories will be performed by applying a tactile stimulation of an application force of 15g (for allodynia) or 0.7g (for hypoesthesia). Tracings will be plotted on tracing paper layer that will then be evaluated by the VISITRAK® tool (Smith & Nephew), validated method reproducible and standardized, enabling accurate measurement of the area concerned .

SUMMARY:
The purpose of this study is to realize a cartography of the allodynic and hypoasthetic territories associated with a neuropathic pain appearing in patients who underwent a Total Knee Arthroplasty (TKA)

DETAILED DESCRIPTION:
The occurrence of Post-surgical Pain depends on the surgical procedure performed, the surgical site and patients-dependents characteristics. Post surgical pain became chronic when it persist beyond two month.

Chronic post-surgical pain (CPSP) is one of the most common complications after surgery. Nerve injury during surgery has been implicated in the development of CPSP. Some patients with CPSP have neuropathic pain (NP). NP is pain cause by damage or disease affecting the somatosensory nervous system. It may be associated with abnormal cutaneous sensation such as hypoesthesia (partial loss of sensitivity to sensory stimuli) or allodynia (pain from normally non-painful stimuli)

Total Knee Arthroplasty (TKA) present a high risk of injury of the infrapatellar branch of the saphenous nerve, thus can cause the appearance of neuropathic post-surgical pain. Only few data are available concerning the skin areas affected after this surgery.

The goal of this study is to analyse the localization of allodynic or hypoasthetic territories that may appear after TKA. The investigators will include 200 patients undergoing TKA surgery at the CHU-Amiens-Picardie. Patient will be seen the day before their surgery, and at follow-up visits at 6 weeks, 6 months and one year postoperatively. A DN diagnostic test (DN4 test) will be performed at each visits. The cartography will be performed on each DN4-positive patients. In addition, patients will also complete questionnaires to assess the intensity of pain, quality of life and level of anxiety.

Thus, the knowledge of the localization of allodynic or hypoasthetic territories will allow a most efficient an faster detection and relief of post-surgical neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* major patient benefit from a first setting operation of TKA (total knee arthroplasty) by standard medial arthrotomy
* Patient signed an informed consent
* Patients receiving social coverage

Exclusion Criteria:

* Patient not wishing to be part of the study, or unable to consent,
* Patient under guardianship or deprived of his liberty
* Patients with neuropathic pain in the territory concerned preoperatively
* Patient who underwent TKA laying by a technique other than standard medial arthrotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patient who received a first setting operation of TKA (total knee arthroplasty)
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Cartography of allodynic and hypoasthetic territories | week 6
  The cartography of allodynic and hypoasthetic territories will be performed by applying a tactile stimulation of an application force of 15g (for allodynia) or 0.7g (for hypoesthesia). Tracings will be plotted on tracing paper layer that will then be evaluated by the VISITRAK® tool (Smith & Nephew), validated method reproducible and standardized, enabling accurate measurement of the area concerned .

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine SORIOT-THOMAS, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France